CLINICAL TRIAL: NCT00496249
Title: The Effect of Radiation on Semen Quality and Fertility in Men Treated With External Beam Radiation or Brachytherapy for Early Stage Prostate Cancer
Brief Title: The Effect of Radiation on Semen Quality and Fertility in Men With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0197-CE
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: Prostate; cancer; brachytherapy; radiation; semen; fertility
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many younger men are diagnosed with prostate cancer. These patients are often choosing radiation therapy as their primary treatment. The effect of this therapy on fertility will have a direct impact on their decision about therapeutic options and fertility preservation. The researchers hypothesize that when patients are treated with radiation for localized prostate cancer, infertility can occur due to direct damage to seminiferous tubules affecting sperm quality.

DETAILED DESCRIPTION:
Prostate cancer is the most common malignant disease among men. Many young men are diagnosed with localized prostate cancer. Some of these men are choosing to manage their prostate cancer with radiation therapy. The radiation therapy delivers minimal dose exposure to adjacent organs. We hypothesize that when patients are treated with radiation therapy for localized prostate cancer, decreased fertility can occur due to damage of seminiferous tubules, which may affect sperm quality. This study will assess the impact of radiation therapy on semen and seminal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed low risk to moderate stage prostate cancer (Gleason 6 - 7) treated with brachytherapy or external beam radiation
* > 12 months ago

Exclusion Criteria:

* Subjects with a prior history of infertility
* Subjects who have undergone vasectomy
* Subjects who have received LHRH therapy for prostate cancer < 6 months ago
* Subjects who have received anti-androgens < 3 months ago
* Subjects using alpha blockers within 7 days of specimen provision
* Subjects who have taken finasteride or dutasteride within the previous 4 months.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men being treated with radiation therapy for localized prostate cancer who consent to participate and provide a semen specimen for analysis following thereapy.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada